CLINICAL TRIAL: NCT04015479
Title: Open-label Randomized Controlled Trial Investigating the Effects of Peanut Protein Powder Supplement on Muscle Growth, Muscle Quality and Other Health Biomarkers in Older Adults Engaging in a Ten-week, Whole-body Resistance Training Program
Brief Title: Peanut Protein Supplementation to Augment Muscle Growth and Improve Markers of Muscle Quality and Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Edward Via Virginia College of Osteopathic Medicine (Other); The Peanut Institute (Other)
Responsible Party: Principal Investigator, Andrew Fruge, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-249
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Aging; Sarcopenia
Keywords: muscle protein synthesis; resistance training; protein supplementation; skeletal muscle physiology; inflammatory cytokines; fecal microbiome; plant protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Intervention group will receive the supplement during the study period and the wait-listed control group will receive the supplement after the study period. Both groups will participate in resistance training during the 10 week period
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI and Co-Is will be blind to participant randomization. One study staff member will be responsible for administering the supplements to participants per randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants will complete 10 weeks of twice-weekly whole body resistance training. Peanut protein powder (72g/day) will be provided for daily consumption during the study period
  Interventions: Dietary Supplement: Peanut Protein Powder; Behavioral: Full body resistance training
- Wait-list Control Group (Active Comparator): Participants will complete 10 weeks of twice-weekly whole body resistance training. Peanut protein powder will be provided after the study period
  Interventions: Behavioral: Full body resistance training

INTERVENTIONS:
Dietary Supplement: Peanut Protein Powder — Peanut protein powder will be provided to participants who will be instructed to consume 72g daily, mixed with water
  Arms: Immediate Intervention Group
Behavioral: Full body resistance training — Participants will undergo supervised resistance training two times per week (5 exercises, 3 sets of 8-12 repetitions per set)

SUMMARY:
This study will evaluate the adaptations in skeletal muscle that occur in response to 10 weeks of weight training with or without peanut protein supplementation in older adult men and women.

DETAILED DESCRIPTION:
Aging is associated with declines in muscle mass, physical strength and physical function. Adequate quality protein intake in aging adults is critical to preventing functional decline. Peanuts provide a unique blend of amino acids that can provide several health benefits to aging adults. While supplementing with peanut protein (PP) powder as part of a resistance training program may increase myofibrillar protein synthesis (i.e., the gold standard molecular assessment in deciphering a muscle-building response), and improve skeletal muscle quality and body composition, no study to date has made this determination.

This is a two-phase study using both novel and conventional methods to assess how PP supplementation affects muscle tissue in older individuals who engage in resistance training. These two phases will be conducted as part of a 10-week randomized controlled trial in which men and women aged 50 years and older (n=60), will be stratified by gender and randomized to a resistance training intervention (whole body, two days per week) with PP powder (72g daily; n=15 males, n=15 females) provided during the intervention (immediate group, IG) or after the intervention (wait-list control, WLC, n=15 males, n=15 females). The aims of this study are to determine the acute (deuterium oxide tracer) and chronic (peripheral quantitative computed tomography) effects of PP during resistance training on skeletal muscle myofibrillar protein synthesis rates, changes in skeletal muscle size and quality, changes in whole and appendicular body composition (dual energy x-ray absorptiometry), changes in inflammatory markers and the fecal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (body mass/height squared) less than 35 kg/m2
* resting blood pressure averaging less than 140/90 mmHg (with or without medication)

Exclusion Criteria:

* known peanut allergy
* actively participating in resistance training for more than 2 days/week
* any known overt cardiovascular or metabolic disease
* metal implants that will interfere with x-ray procedures
* medically necessary radiation exposure in the last six months (except dental x-ray)
* any medical condition that would contradict participating in an exercise program, giving blood or donating a skeletal muscle biopsy (i.e. blood clotting disorder or taking blood thinners)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in acute myofibrillar protein synthesis rates | 24 hours
  Change in right leg vastus lateralis myofibrillar protein synthesis rates using the integrated deuterium oxide technique from biopsies immediately before and 24 hours after resistance exercise
Change in mid-thigh skeletal muscle area and quality | 0-10 weeks
  peripheral quantitative computed tomography (pQCT) cross-sectional image of mid-right thigh assessed for total muscle cross-sectional area, subcutaneous adipose tissue area, total intra- and inter-muscular adipose tissue area and overall muscle density

SECONDARY OUTCOMES:
Change in whole-body and appendicular body composition | 0-10 weeks
  dual energy x-ray absorptiometry (DXA)
Change in Type I and II Muscle Fiber Cross-Sectional Area | 0-10 weeks
  Muscle biopsy immunofluorescent staining for determination of type I and type II muscle fiber cross sectional area (fCSA) as a cellular determinant of skeletal muscle hypertrophy
Change in leg extensor isokinetic dynamometry | 0-10 weeks
  maximal isokinetic right leg extensions on an isokinetic dynamometer (BioDex)
Change in inflammatory biomarkers | 0-10 weeks
  serum C-reactive protein, interleukin-6, tumor necrosis factor-alpha, plasma 8-hydroxy-2'deoxyguanosine
Change in fecal microbiome composition | 0-10 weeks
  alpha- and beta-diversity of 16S bacterial rDNA

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roberts, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

REFERENCES:
- [Background] Lamb DA, Moore JH, Smith MA, Vann CG, Osburn SC, Ruple BA, Fox CD, Smith KS, Altonji OM, Power ZM, Cerovsky AE, Ross CO, Cao AT, Goodlett MD, Huggins KW, Fruge AD, Young KC, Roberts MD. The effects of resistance training with or without peanut protein supplementation on skeletal muscle and strength adaptations in older individuals. J Int Soc Sports Nutr. 2020 Dec 14;17(1):66. doi: 10.1186/s12970-020-00397-y. PMID 33317565